CLINICAL TRIAL: NCT02420041
Title: Comparison of the Efficacy of Two Techniques for Sacroiliac Joint Injection: Ultrasound Guidance Versus Fluoroscopic Guidance
Brief Title: Comparing the Effects of Ultrasound Versus Fluoroscopy for Sacroiliac Joint Injections
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: United States Naval Medical Center, San Diego (U.S. Federal Agency)
Collaborators: United States Naval Medical Center, Portsmouth (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NMCSD.2012.0112
Record Dates: First submitted 2014-09-30; First posted 2015-04-17 (Estimated); Results first posted 2015-11-13 (Estimated); Last update posted 2015-11-13 (Estimated); Status verified 2015-10

CONDITIONS: Sacroiliitis
Keywords: Sacroiliac Joint Injection; Fluoroscopy; Ultrasound
MeSH Terms: conditions — Sacroiliitis | interventions — Triamcinolone; Lidocaine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Fluoroscopic Guidance (Active Comparator): Patients referred to the Naval Medical Center-San Diego Pain Medicine Clinic. Need a history and physical showing objective findings of sacroiliac joint (SIJ) dysfunction. If the patient meets inclusion / exclusion criteria, they will be presented with the study. After accepting and being consented, they will then be scheduled. The day of the appointment they will be randomised to Group A or B. In Group A : Fluoroscopy will be used to Guide Needle Placement to inject Steroid into joint. Then complete the multidimensional pain inventory (MPI) and rate their pain on the NRS from 0-11. After procedure, they will rate their pain from 0-10 in the recovery area and then be discharged to home. They will complete an MPI, Patient Global Impression of Change (PGIC), numerical rating scale (NRS), and adverse events questionnaire 1-2 weeks post-procedure and 3 months post-procedure.
  Interventions: Procedure: Active comparator: Fluoroscopic Guided SIJ injection; Device: Havel's Inc. EchoStim (facet tip) 21 Gauge 4" needle; Device: iohexol; Drug: triamcinolone/lidocaine
- Ultrasound Guidance (Experimental): Patients referred to the Naval Medical Center-San Diego Pain Medicine Clinic. Need a history and physical showing objective findings of SIJ dysfunction. If the patient meets inclusion / exclusion criteria, they will be presented with the study. After accepting and being consented, they will then be scheduled. The day of the appointment they will be randomised to Group A or B. In Group B Ultrasound will be used to Guide Needle Placement to inject steroid into joint. Then complete the MPI and rate their pain on the NRS from 0-11. After procedure, they will rate their pain from 0-10 in the recovery area and then be discharged to home. They will complete an MPI, Patient Global Impression of Change (PIGC), NRS, and adverse events questionnaire 1-2 weeks post-procedure and 3 months post-procedure.
  Interventions: Procedure: Ultrasound Guided Sacroiliac Joint Injection; Device: Havel's Inc. EchoStim (facet tip) 21 Gauge 4" needle; Device: SonoSite S-nerve; Drug: triamcinolone/lidocaine

INTERVENTIONS:
Procedure: Active comparator: Fluoroscopic Guided SIJ injection — * Needle entry point is in the lower one-third of the SIJ
  * Sterile preparation (with chlorhexidine) and draping and 3 mL of 1% lidocaine injected subcutaneously at site of needle entry
  * Under fluoroscopy guidance, Havel's Inc. EchoStim (facet tip) 21 Gauge 4" needle is inserted in a coaxial fashion into the SIJ
  * 1 mL of contrast (iohexol 300 mg/mL) is injected to outline the SIJ and to ensure no vascular uptake
  * Injection of 20 mg of triamcinolone diluted in 4 mL of 1% lidocaine
  * Patient observed in recovery bay for 20 minutes and then discharged home
  Arms: Fluoroscopic Guidance
Procedure: Ultrasound Guided Sacroiliac Joint Injection — * Sterile preparation (with chlorhexidine) and drape
  * Using ultrasound guidance (SonoSite S-nerve) with a low frequency (2-5 Hz) curvilinear transducer in a sterile cover, the transducer is placed in a transverse plane over the SIJ and needle entry point is chosen at the medial end of the ultrasound transducer
  * 3 mL of 1% lidocaine is injected subcutaneously at site of needle entry
  * Under ultrasound guidance, a Havel's Inc. EchoStim (facet tip) 21 Gauge 4" needle is inserted in a medial to lateral direction and guided into the SIJ. (0.5-2 mL of normal saline may be injected during needle insertion to locate tip of needle and to ensure solution does not "spill out" onto sacrum).
  * After using the Doppler function to identify any surrounding vessels (to avoid intravascular injection), 20 mg of triamcinolone diluted in 4 mL of 1% lidocaine is injected.
  * Patient observed in recovery bay for 20 minutes and then discharged home
  Arms: Ultrasound Guidance
Device: Havel's Inc. EchoStim (facet tip) 21 Gauge 4" needle
Device: SonoSite S-nerve
  Arms: Ultrasound Guidance
Device: iohexol
  Arms: Fluoroscopic Guidance
Drug: triamcinolone/lidocaine

SUMMARY:
The purpose of this research project is to compare two different techniques for performing an injection of the sacroiliac joint. Although both techniques are safe and accurate, the goal of the study is to determine if one technique is better than the other with respect to improvement in a patient's pain, function, and his or her satisfaction. Additionally, the investigators want to determine if one technique is quicker and more efficient than the other.

DETAILED DESCRIPTION:
Sacroiliac joint dysfunction is a source of low back pain that causes significant pain and disability. Injection of the sacroiliac joint with a local anesthetic/corticosteroid mixture has shown efficacy in treating this condition, when conservative therapy fails. The use of fluoroscopic guidance and anatomic landmarks are traditional methods for performing this injection; however, ultrasound imaging has recently been utilized for performing this procedure. Although studies exist that describe and validate the ultrasound technique, no studies exist that compare the techniques with respect to short-term and long-term outcomes. In this study, the primary objective is to determine if a difference exists between a fluoroscopic-guided technique and ultrasound-guided technique with respect to pain and function. A secondary objective is to compare the two techniques with respect to procedural characteristics.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of SIJ dysfunction by history and physical exam

   * History: Either low back pain or buttock pain
   * Exam: Either tenderness to palpation over the SIJ or a positive provocative maneuver (i.e., Patrick's, Gaenslen's, and/or Yeoman's test)
2. Failed a trial of conservative therapy which may included medications, physical therapy, or both
3. Age > 18
4. Patient agrees to participate in study

Exclusion Criteria:

1. Coagulopathy
2. Renal or Hepatic Failure
3. Current Pregnancy or actively pursuing pregnancy
4. Known allergy to local anesthetic or steroids
5. Infection at site of needle placement or SIJ infection
6. Patient unable to consent himself or herself
7. Patient refusal
8. Prior surgical procedures involving the SIJ
9. Body Mass Index > 35 kg/m2

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2012-10; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven R Hanling, MD, Principal Investigator — United States Naval Medical Center, San Diego
Locations (1):
- Pain Medicine Center, Department of Anesthesiology, Naval Medical Center, San Diego, San Diego, California, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Fluoroscopic Guidance: In Group A : Fluoroscopy will be used to Guide Needle Placement to inject Steroid into joint.
  * Needle entry point is in the lower one-third of the sacroiliac joint (SIJ)
  * Under fluoroscopic guidance, Havel's Inc. EchoStim 21 gauge 4" needle is inserted in a coaxial fashion into the SIJ
- Ultrasound Guidance: In Group B Ultrasound will be used to Guide Needle Placement to inject steroid into joint.
  * Using ultrasound guidance (SonoSite S-nerve) with a low frequency (2-5 Hz) curvilinear transducer in a sterile cover, the transducer is placed in a transverse plane over the SIJ and needle entry point is chosen at the medial end of the ultrasound transducer.
  * Under ultrasound guidance, a Havel's Inc. EchoStim 21 gauge 4" needle is inserted in a medial to lateral direction and guided into the SIJ.
Period: Overall Study
Arm/Group | Fluoroscopic Guidance | Ultrasound Guidance
Started | 14 | 14
Completed | 14 | 14
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Fluoroscopic Guidance: In Group A : Fluoroscopy will be used to Guide Needle Placement to inject Steroid into joint.
  * Needle entry point is in the lower one-third of the SIJ
  * Under fluoroscopic guidance, Havel's Inc. EchoStim 21 gauge 4" needle is inserted in a coaxial fashion into the SIJ
- Total: Total of all reporting groups
Arm/Group | Fluoroscopic Guidance | Ultrasound Guidance | Total
Number analyzed (Participants) | 14 | 14 | 28
Age, Continuous [Mean (Standard Deviation); unit: years] | 37 (7.6175) | 34.07 (8.2695) | 35.535 (7.9435)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 5 | 11
  Male | 8 | 9 | 17
Region of Enrollment [Number; unit: participants]
  United States | 14 | 14 | 28

OUTCOME MEASURES:

1. Primary Outcome: Difference in Minutes Between a Sacroiliac Joint Injection Done With Ultrasound vs Fluoroscopy
Description: during procedure from the time monitors are placed on patient to the time of withdrawal of needle from skin
Time Frame: difference in minutes between a sacroiliac joint injection, an expected average of 9 minutes
Measure: Mean (Full Range); unit: minutes
Arm/Group | Fluoroscopic Guidance | Ultrasound Guidance
Number analyzed (Participants) | 14 | 14
minutes | 9.471 [6.92 to 15] | 9.552 [3 to 30]

2. Primary Outcome: Change in Pain Score From Baseline to 30 Minutes Pre-procedure Using the Defense and Veterans Pain Rating Scale (DoD/VA PRS) 0-10
Description: Study subjects rate their pain on a scale of 0-10 (0=no pain, 10= the highest level of pain experienced), hence the lower the score the better the outcome.
Time Frame: 30 minutes pre-procedure minus baseline
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Fluoroscopic Guidance | Ultrasound Guidance
Number analyzed (Participants) | 14 | 14
units on a scale | -2.571 [-5 to 0] | -2.571 [-7 to 0]

3. Primary Outcome: Change in Pain Score From Baseline to 2 Weeks Post-procedure Using the DoD/VA PRS
Description: as for outcome 2
Time Frame: 2 weeks post-procedure minus baseline
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Fluoroscopic Guidance | Ultrasound Guidance
Number analyzed (Participants) | 14 | 14
units on a scale | -1 [-3 to 0] | -1.643 [-6 to 0]

4. Primary Outcome: Change in Pain Score From Baseline to 3 Months Post-procedure Using the DoD/VA PRS
Description: as for outcome 2
Time Frame: 3 months post-procedure minus baseline
Population: numbers of participants analyzed are not consistent because study subjects were lost to follow-up along different points in time in the study
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Fluoroscopic Guidance | Ultrasound Guidance
Number analyzed (Participants) | 12 | 9
units on a scale | -0.875 [-2 to .5] | -1.556 [-5 to 0]

5. Secondary Outcome: Impression of Change of Condition at 2 Weeks Post-procedure Using the Patient Global Impression of Change (PGIC) Scale
Description: Study subjects rate their change in overall condition on a scale of 0-6 (0=no change, 6=better and a definite improvement that has made a real worthwhile difference). The range of the change in pain for both groups observed was in fact 0-5.
Time Frame: 2 weeks post-procedure
Population: as for outcome 4
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Fluoroscopic Guidance | Ultrasound Guidance
Number analyzed (Participants) | 13 | 14
units on a scale | 2.385 [0 to 5] | 2.714 [0 to 5]

6. Secondary Outcome: Impression of Change of Condition at 3 Months Post-procedure Using the PGIC Scale
Description: as for outcome 5
Time Frame: 3 months post-procedure
Population: as for outcome 4
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Fluoroscopic Guidance | Ultrasound Guidance
Number analyzed (Participants) | 11 | 9
units on a scale | 2.818 [0 to 5] | 2.222 [0 to 5]

7. Secondary Outcome: Change in Pain Score Since Sacroiliac (SI) Injection at 2 Weeks Post-procedure Using the DoD/VA PRS
Description: Study subjects rate their pain on a scale of 0-10 (0=no pain, 10= the highest level of pain experienced), hence the lower the score the better the outcome. Score reported is reporting a difference/change between two time points.
Time Frame: during/just before sacroiliac (SI) injection and 2 weeks post-procedure
Population: as for outcome 4
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Fluoroscopic Guidance | Ultrasound Guidance
Number analyzed (Participants) | 13 | 13
units on a scale | 4.846 [0 to 8] | 4.385 [2 to 9]

8. Secondary Outcome: Change in Pain Score Since SI Injection at 3 Months Post-procedure Using the DoD/VA PRS
Description: Study subjects rate their pain on a scale of 0-10 (0=no pain, 10= the highest level of pain experienced), hence the lower the score the better the outcome.Score reported is reporting a difference/change between two time points.
Time Frame: during/just before sacroiliac (SI) injection and 3 months post-procedure
Population: as for outcome 4
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Fluoroscopic Guidance | Ultrasound Guidance
Number analyzed (Participants) | 10 | 9
units on a scale | 4 [1 to 7] | 4.333 [3 to 8]

9. Secondary Outcome: Satisfaction of Procedure as a Measure of Safety and Tolerability Using a Numerical Scale 1-5
Description: "1= very dissatisfied" to "5=very satisfied".
Time Frame: 2 weeks post-procedure
Population: as for outcome 4
Measure: Mean (Full Range); unit: units on a scale of satisfaction
Arm/Group | Fluoroscopic Guidance | Ultrasound Guidance
Number analyzed (Participants) | 13 | 14
units on a scale of satisfaction | 3.615 [1 to 5] | 3.857 [2 to 5]

10. Secondary Outcome: Satisfaction of Procedure as a Measure of Safety and Tolerability Using a Numerical Scale 1-5
Description: "1= very dissatisfied" to "5=very satisfied".
Time Frame: 3 months post-procedure
Population: as for outcome 4
Measure: Mean (Full Range); unit: units on a scale of satisfaction
Arm/Group | Fluoroscopic Guidance | Ultrasound Guidance
Number analyzed (Participants) | 11 | 9
units on a scale of satisfaction | 3.364 [2 to 4] | 3.667 [3 to 4]

ADVERSE EVENTS:
Description: All adverse events, including serious adverse events, were collected but none occurred. Data input includes all non-serious adverse events that occurred during this study.
Arm/Group | Fluoroscopic Guidance | Ultrasound Guidance
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/14
Other Adverse Events (participants affected / at risk) | 5/14 | 3/14
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fluoroscopic Guidance (N=14) | Ultrasound Guidance (N=14)
Vasovagal reaction (Cardiac disorders) | 1 (1) | 1 (1)
Facetogenic back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Lower back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Myofascial pain syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Sacroiliac joint pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes